CLINICAL TRIAL: NCT03585946
Title: A Prospective Multicenter Cohort Study Assessing Outcomes in Stevens Johnsons Syndrome and Toxic Epidermal Necrolysis
Brief Title: Outcomes in Stevens Johnsons Syndrome and Toxic Epidermal Necrolysis
Status: Withdrawn | Type: Observational
Why Stopped: Change in study design
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniela Kroshinsky, Associate Professor of Dermatology, Massachusetts General Hospital
Other Study IDs: P201700P002792
Record Dates: First submitted 2018-03-14; First posted 2018-07-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stevens-Johnson Syndrome; Toxic Epidermal Necrolysis; Drug Reaction
MeSH Terms: conditions — Stevens-Johnson Syndrome; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Cyclosporine
  Interventions: Drug: Site specific standard of care comparison
- Intravenous Immunoglobulin
  Interventions: Drug: Site specific standard of care comparison
- Etanercept
  Interventions: Drug: Site specific standard of care comparison
- Steroids
  Interventions: Drug: Site specific standard of care comparison

INTERVENTIONS:
Drug: Site specific standard of care comparison — Patients outcomes will be assessed and compared based on the medication they receive which will be assigned based on the standard of care at each enrolling site.

SUMMARY:
This is a prospective, multicenter cohort observational; study to compare treatment outcomes in patients admitted to the hospital with Stevens-Johnsons Syndrome/Toxic Epidermolysis, aiming to assess the utility of medical management. The hypothesis of this study is that one or more treatment options will demonstrate improved patient outcomes. The primary objectives are cessation of progression of disease, time to complete re-epithelialization, length of stay, and mortality rate in the treatment groups as compared to those receiving supportive care alone. Exploratory analyses will assess the cause, risk factors, and severity prediction factors associated with the disease.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of Stevens Johnsons Syndrome/Toxic Epidermal Necrolysis confirmed by examination of a dermatologist and/or skin biopsy plus described appropriate clinical findings (epidermal necrosis plus two involved mucosal surfaces) presenting within one week of disease onset

Exclusion Criteria:

* Pregnancy
* Age <18y
* Decisional impairment
* Incarceration
* Onset of skin separation >7d

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized with a diagnosis of Stevens Johnsons Syndrome/Toxic Epidermal Necrolysis confirmed by examination of a dermatologist and/or skin biopsy plus described appropriate clinical findings (epidermal necrosis plus two involved mucosal surfaces) presenting within one week of disease onset.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2030-01-01 (Estimated); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 years
  Percent of deaths in each group
Time to cessation of new lesion formation | 3 years
  Days until no new lesions arise from time of initiation of therapy
Time to re-epithelialization | 3 years
  Days until skin has completely healed
Hospital length of stay | 3 years
  Time from hospital admission to discharge

IPD SHARING:
Plan to Share IPD: Yes
Data to be recorded includes age, gender, past medical history, medications prior to admission, allergies, physical exam including body sites and surface area involved, pain scores, laboratory values, imaging results, and outcome in terms of morbidity and mortality. The privacy of subjects and their data will be maintained by de-identifying patient data by substituting codes for medical record numbers.
Supporting Information: Study Protocol, SAP, ICF, CSR